CLINICAL TRIAL: NCT05893862
Title: A Double-Blind, Cross-Over Placebo-Controlled and Active-Controlled Trial To Evaluate The Effect Of A Supratherapeutic Dose Of MK-8189 On The QTc Interval In Participants With Schizophrenia
Brief Title: A Study To Evaluate The Effect Of A Supratherapeutic Dose Of MK-8189 On The QTc Interval In Participants With Schizophrenia (MK-8189-019)
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8189-019; MK-8189-019 (Other: Merck)
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1: MK-8189 (Treatment A)→Moxifloxacin (Treatment B)→Placebo (Treatment C) (Experimental): Participants receive a sequence of Treatment A in Period 1 followed by Treatment B in Period 2 followed by Treatment C in Period 3; there will be a 5-day washout between periods. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on day 2. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2. Treatment C consists of placebo administered orally on Day 1 and Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo
- Sequence 2: Moxifloxacin (Treatment B) →Placebo (Treatment C) →MK-8189 (Treatment A) (Experimental): Participants receive a sequence of Treatment B in Period 1 followed by Treatment C in Period 2 followed by Treatment A in Period 3; there will be a 5-day washout between periods. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2. Treatment C consists of placebo administered orally on Day 1 and Day 2. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo
- Sequence 3: Placebo (Treatment C) →MK-8189 (Treatment A) →Moxifloxacin (Treatment B) (Experimental): Participants receive a sequence of Treatment C in Period 1 followed by Treatment A in in Period 2 followed by Treatment B in Period 3; there will be a 5-day washout between periods. Treatment C consists of placebo administered orally on Day 1 and Day 2. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on Day 2. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo
- Sequence 4: Moxifloxacin (Treatment B) → MK-8189 (Treatment A) → Placebo (Treatment C) (Experimental): Participants receive a sequence of Treatment B in Period 1 followed by Treatment A in Period 2 followed by Treatment C in Period 3; there will be a 5-day washout between periods. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on Day 2. Treatment C consists of placebo administered orally on Day 1 and Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo
- Sequence 5: MK-8189 (Treatment A) →Placebo (Treatment C) →Moxifloxacin (Treatment B) (Experimental): Participants receive a sequence of Treatment A in Period 1 followed by Treatment C in Period 2 followed by Treatment B in Period 3; there will be a 5-day washout between periods. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on Day 2. Treatment C consists of placebo administered orally on Day 1 and Day 2. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo
- Sequence 6: Placebo (Treatment C) →Moxifloxacin (Treatment B) → MK-8189 (Treatment A) (Experimental): Participants receive a sequence of Treatment C in Period 1 followed by Treatment B in Period 2 followed by Treatment A in Period 3; there will be a 5-day washout between periods. Treatment C consists of placebo administered orally on Day 1 and Day 2. Treatment B consists of placebo administered orally on Day 1 and moxifloxacin administered orally at 400 mg on Day 2. Treatment A consists of MK-8189 administered orally at 48 mg on Day 1 and 80 mg on Day 2.
  Interventions: Drug: MK-8189; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — Oral Tablet
Drug: Moxifloxacin — Oral Tablet
Drug: Placebo — Oral Tablet

SUMMARY:
The primary purpose of this study to evaluate the effect of a supratherapeutic dose of 80 mg MK-8189 on the QT interval corrected for heart rate (QTc interval) and to assess the safety and tolerability of multiple once-daily doses of MK-8189 in participants with schizophrenia. The effects of 3 treatment sequences 1) MK-8189 (48 mg [Day 1] and 80 mg [Day2]); 2) standard image placebo (Day 1) and moxifloxacin 400 mg (Day 2); and 3) MK-8189 placebo (Day 1 and Day 2) were assessed with 5-day washout intervening sequence. Participants received all treatments in a counter-balanced order according to 1 of 6 possible treatment sequences.

The primary hypothesis is that the administration of an 80 mg MK-8189 dose on Day 2 does not prolong the QTc interval to a clinically significant degree. Specifically, the true mean difference (MK-8189 - placebo) in QTc change from baseline is less than 10 milliseconds (msec).

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.
* Is in the non-acute phase of their illness.
* Has a history of receiving and tolerating antipsychotics medication within the usual dose range employed for schizophrenia.
* Participants with hypothyroidism, diabetes, high blood pressure, chronic respiratory conditions or other medical conditions could be considered if their condition is stable.

Exclusion Criteria:

* History of a primary DSM-5 axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder per the allowed DSM-5 criteria.
* History of intellectual disability, borderline personality disorder, anxiety disorder, or organic brain syndrome.
* History of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia (TD).
* History of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures.
* History of cancer.
* History or presence of sick sinus syndrome, atrioventricular (AV) block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QTc interval, or conduction abnormalities.
* History of risk factors for Torsades de Pointes (e.g., heart failure/cardiomyopathy or family history of long QT syndrome).
* History of frequent syncope, vasovagal episodes, or epileptic seizures.
* Family history of sudden cardiac death.
* Has a positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated, or lost 1 unit of blood within 4 weeks prior to the pre-study visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - California Clinical Trials Medical Group managed by PAREXEL-PAREXEL International ( Site 0003), Glendale, California
  - NRC Research Institute ( Site 0004), Orange, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0002), Hallandale, Florida
  - Hassman Research Institute Marlton Site ( Site 0001), Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with stable schizophrenia or schizoaffective disorder were enrolled at 4 study sites in the US.
Pre-assignment Details: Treatments were administered in a counterbalanced manner on Day 1 and Day 2 of each of 3 treatment periods. Periods 1 and 2 were separated by 5-day washout. 'A' refers to MK-8189 48 mg (Day 1) and 80 mg (Day 2); 'B' refers to Standard Image Placebo (Day 1) and Moxifloxacin 400 mg (Day 2); and 'C' refers to placebo to MK-8189 (Days 1 and 2).
Groups:
- Sequence A/B/C: Participants received treatment sequence A/B/C.
- Sequence A/C/B: Participants received treatment sequence A/C/B.
- Sequence B/A/C: Participants received treatment sequence B/A/C.
- Sequence B/C/A: Participants received treatment sequence B/C/A.
- Sequence C/A/B: Participants received treatment sequence C/A/B.
- Sequence C/B/A: Participants received treatment sequence C/B/A.
Period: Overall Study
Arm/Group | Sequence A/B/C | Sequence A/C/B | Sequence B/A/C | Sequence B/C/A | Sequence C/A/B | Sequence C/B/A
Started (Randomized) | 15 | 25 | 15 | 18 | 20 | 14
Treatment Period 1 + 5 Day Washout | 15 | 25 | 15 | 18 | 20 | 14
Treatment Period 2 + 5 Day Washout | 14 | 16 | 15 | 15 | 18 | 14
Treatment Period 3 | 13 | 13 | 12 | 13 | 15 | 12
Completed | 13 | 13 | 12 | 13 | 15 | 12
Not Completed | 2 | 12 | 3 | 5 | 5 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 7 | 1 | 3 | 3 | 2
Not completed — Adverse Event | 1 | 4 | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence ACB: Participants received treatment sequence A/C/B.
- Total: Total of all reporting groups
Arm/Group | Sequence A/B/C | Sequence ACB | Sequence B/A/C | Sequence B/C/A | Sequence C/A/B | Sequence C/B/A | Total
Number analyzed (Participants) | 15 | 25 | 15 | 18 | 20 | 14 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.3) | 46.0 (10.9) | 43.5 (9.8) | 46.8 (7.6) | 44.1 (9.3) | 45.9 (11.2) | 45.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 3 | 4 | 3 | 3 | 24
  Male | 12 | 17 | 12 | 14 | 17 | 11 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4 | 2 | 3 | 13
  Not Hispanic or Latino | 14 | 23 | 14 | 14 | 18 | 11 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 12 | 21 | 13 | 14 | 17 | 9 | 86
  White | 3 | 3 | 2 | 2 | 1 | 5 | 16
  More than one race | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in QT Interval Corrected for Heart Rate (QTc) Following Moxifloxacin Treatment
Description: Electrocardiogram data was obtained using a digital Holter device and the Fridericia correction of the QT interval (QTcF) was determined. The change from baseline in QTcF (ΔQTcF [msec]) was calculated by subtracting the QTcF value at the timepoint from the QTcF baseline value. Negative values represent a decrease from baseline and vice versa. An average of up to 9 predose ECGs on Day 1 served as baseline to compare postdose effects. Per protocol, the secondary endpoint compares moxifloxacin to placebo on Day 2. Moxifloxacin was tested for statistical significance 1 to 4 hours postdose (ie, around moxifloxacin Cmax) to ensure assay sensitivity. Hochberg's step-up method was applied to preserve the overall α level at .05 for the hypothesis testing.
Time Frame: Day 2
Population: All participants who received ≥1 dose of moxifloxacin, and who complied with the protocol sufficiently to ensure that generated data will likely exhibit the effects of treatment (according to the underlying scientific model), are included.
Measure: Mean (95% Confidence Interval); unit: ΔQTcF (msec)
Groups:
- MK-8189 48 mg Day 1: Participants received a single dose of MK-8189 48 mg.
- Placebo Day 1; Placebo Day 2: Participants received a single dose of placebo.
- MK-8189 80 mg Day 2: Participants received a single dose of MK-8189 80 mg.
- Standard Image Placebo Day 1: Participants received a single dose of standard image placebo on Day 1.
- Moxifloxacin 400 mg Day 2: Participants received a single dose of moxifloxacin 400 mg on Day 2. Standard image placebo was given on Day 1 (open-label).
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 0 | 0 | 0 | 84 | 0 | 84
ΔQTcF (msec)
  Predose (Day 2 only) |  |  |  | -1.38 [-3.24 to 0.49] |  | 0.92 [-0.80 to 2.65]
  0.5 hr (Day 1 only): number analyzed (Participants) | 0 | 0 | 0 | 84 | 0 | 0
  0.5 hr (Day 1 only) |  |  |  | -1.38 [-3.24 to 0.49] |  |
  1 hr: number analyzed (Participants) | 0 | 0 | 0 | 82 | 0 | 83
  1 hr |  |  |  | -0.76 [-2.95 to 1.43] |  | 9.77 [7.34 to 12.20]
  2 hr: number analyzed (Participants) | 0 | 0 | 0 | 83 | 0 | 81
  2 hr |  |  |  | 0.92 [-1.74 to 3.58] |  | 11.03 [8.53 to 13.53]
  3 hr: number analyzed (Participants) | 0 | 0 | 0 | 82 | 0 | 81
  3 hr |  |  |  | -2.22 [-5.17 to 0.72] |  | 8.92 [6.28 to 11.57]
  4 hr: number analyzed (Participants) | 0 | 0 | 0 | 83 | 0 | 82
  4 hr |  |  |  | -2.67 [-5.40 to 0.05] |  | 4.70 [1.84 to 7.57]
  8 hr: number analyzed (Participants) | 0 | 0 | 0 | 84 | 0 | 82
  8 hr |  |  |  | -3.10 [-5.82 to -0.39] |  | 3.50 [1.05 to 5.95]
  11 hr: number analyzed (Participants) | 0 | 0 | 0 | 84 | 0 | 83
  11 hr |  |  |  | -1.93 [-4.83 to 0.98] |  | 5.45 [2.85 to 8.04]
  14 hr: number analyzed (Participants) | 0 | 0 | 0 | 83 | 0 | 81
  14 hr |  |  |  | 0.84 [-2.54 to 4.22] |  | 10.12 [6.90 to 13.35]
  16 hr: number analyzed (Participants) | 0 | 0 | 0 | 83 | 0 | 82
  16 hr |  |  |  | 5.20 [2.23 to 8.17] |  | 12.48 [9.37 to 15.59]
  24 hr: number analyzed (Participants) | 0 | 0 | 0 | 84 | 0 | 73
  24 hr |  |  |  | -.61 [-3.22 to -0.01] |  | 2.33 [-0.08 to 4.74]
Statistical Analysis 1: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 1 Hr; p < 0.0001, t-test, 1 sided; LS Mean Difference = 9.22, 90% CI 2-sided [7.40 to 11.04]
Statistical Analysis 2: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 2 Hr; p = 0.0141, t-test, 1 sided; LS Mean Difference = 8.44, 90% CI 2-sided [6.31 to 10.56]
Statistical Analysis 3: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 3 Hr; p < 0.0001, t-test, 1 sided; LS Mean Difference = 10.80, 90% CI 2-sided [8.85 to 12.74]
Statistical Analysis 4: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference Week 4 Hr; p = 0.1045, t-test, 1 sided; LS Mean Difference = 6.43, 90% CI 2-sided [3.96 to 8.91]
Statistical Analysis 5: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 8 Hr; LS Mean Difference = 6.52, 90% CI 2-sided [4.66 to 8.38]
Statistical Analysis 6: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 11 Hr; LS Mean Difference = 7.33, 90% CI [4.74 to 9.93]
Statistical Analysis 7: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 14 Hr; LS Mean Difference = 6.42, 90% CI 2-sided [3.95 to 8.88]
Statistical Analysis 8: Comparison: Placebo Day 2 vs Moxifloxacin 400 mg Day 2; Test type: Other — LS Mean Difference 24 Hr; LS Mean Difference = 2.79, 90% CI 2-sided [0.81 to 4.76]

2. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of MK-8189
Description: AUC0-24 is defined as the area under concentration-time curve from 0 to 24 hours postdose. Blood samples taken at pre-dose and up to 24 hours post-dose will be used to determine the AUC0-24 of MK-8189.
Time Frame: Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24 hours postdose; Day 2: 0.5, 1, 2, 3, 4, 8, 11, 14, 16, 24 hours postdose
Population: All participants who received ≥1 dose of MK-8189, and who complied with the protocol sufficiently to ensure that generated data will likely exhibit the effects of treatment (according to the underlying scientific model), are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Groups:
- Standard Image Placebo Day 1: Participants received a single dose of placebo.
- Moxifloxacin 400 mg Day 2: Participants received a single dose of moxifloxacin 400 mg.
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 91 | 0 | 87 | 0 | 0 | 0
hr*nM | 18500 (50.2) |  | 41200 (54.0) |  |  |

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of MK-8189
Description: AUC0-last is defined as the area under concentration-time curve from 0 to 24 hours. Blood samples taken at pre-dose and up to 72 hours post-dose will be used to extrapolate the AUC0-last of MK-8189.
Time Frame: Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24 hours postdose; Day 2: 0.5, 1, 2, 3, 4, 8, 11, 14, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 96 | 0 | 91 | 0 | 0 | 0
hr*nM | 17400 (61.6) |  | 54100 (95.9) |  |  |

4. Primary Outcome: Change From Baseline in QT Interval Corrected for Heart Rate (QTc) Following MK-8189 Treatment
Description: Electrocardiogram data was obtained using a digital Holter device and the Fridericia correction of the QT interval (QTcF) was determined. The change from baseline in QTcF (ΔQTcF [msec]) was calculated by subtracting the QTcF value at the timepoint from the QTcF baseline value. Negative values represent a decrease from baseline and vice versa. An average of up to 9 predose ECGs on Day 1 served as baseline to compare postdose effects. Per protocol, the primary endpoint compares MK-8189 to placebo.
Time Frame: Day 1 (MK-8189 48 mg and placebo) and Day 2 (MK-8189 80 mg and placebo)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ΔQTcF (msec)
Groups:
- Moxifloxacin 400 mg Day 2: Participants received a single dose of moxifloxacin 400 mg on Day 2.
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 95 | 87 | 91 | 84 | 0 | 0
ΔQTcF (msec)
  Predose (Day 2 only): number analyzed (Participants) | 0 | 0 | 89 | 84 | 0 | 0
  Predose (Day 2 only) |  |  | 4.31 [2.45 to 6.16] | -1.38 [-3.24 to 0.49] |  |
  0.5 Hr: number analyzed (Participants) | 95 | 86 | 0 | 0 | 0 | 0
  0.5 Hr | -0.61 [-1.87 to 0.66] | -1.13 [-2.84 to 0.57] |  |  |  |
  1 hr: number analyzed (Participants) | 95 | 83 | 90 | 80 | 0 | 0
  1 hr | 0.29 [-1.50 to 2.08] | 0.48 [-1.25 to 2.20] | 3.60 [1.33 to 5.87] | -0.76 [-2.95 to 1.43] |  |
  2 hr: number analyzed (Participants) | 94 | 86 | 91 | 82 | 0 | 0
  2 hr | 2.68 [0.21 to 5.16] | 1.06 [-1.35 to 3.46] | 5.14 [2.40 to 7.87] | 0.92 [-1.74 to 3.58] |  |
  3 hr: number analyzed (Participants) | 94 | 87 | 89 | 81 | 0 | 0
  3 hr | 2.18 [-0.61 to 4.97] | -1.35 [-4.03 to 1.34] | 3.31 [0.50 to 6.11] | -2.22 [-5.17 to 0.72] |  |
  4 hr: number analyzed (Participants) | 95 | 84 | 87 | 83 | 0 | 0
  4 hr | 2.80 [0.07 to 5.53] | -3.19 [-5.73 to -0.64] | 2.64 [0.11 to 5.16] | -2.67 [-5.40 to 0.05] |  |
  6 hr (Day 1 only): number analyzed (Participants) | 93 | 85 | 0 | 82 | 0 | 0
  6 hr (Day 1 only) | 7.38 [4.75 to 10.00] | 0.25 [-2.51 to 3.02] |  | -3.10 [-5.82 to -0.39] |  |
  8 hr: number analyzed (Participants) | 89 | 85 | 84 | 81 | 0 | 0
  8 hr | 8.75 [6.51 to 10.98] | -0.97 [-3.57 to 1.64] | 2.82 [0.25 to 5.40] | -1.93 [-4.83 to 0.98] |  |
  12 hr (Day 1) or 11 hr (Day 2): number analyzed (Participants) | 89 | 84 | 89 | 79 | 0 | 0
  12 hr (Day 1) or 11 hr (Day 2) | 4.26 [1.41 to 7.11] | 0.33 [-2.12 to 2.79] | 3.84 [0.95 to 6.73] | 0.84 [-2.54 to 4.22] |  |
  14 hr: number analyzed (Participants) | 90 | 84 | 86 | 79 | 0 | 0
  14 hr | 8.10 [5.33 to 10.86] | 4.09 [1.66 to 6.53] | 7.84 [7.53 to 13.42] | 5.20 [2.23 to 8.17] |  |
  16 hr (Day 2 only): number analyzed (Participants) | 0 | 0 | 83 | 80 | 0 | 0
  16 hr (Day 2 only) |  |  | 10.47 [7.53 to 13.42] | 5.20 [2.23 to 8.17] |  |
  24 hr: number analyzed (Participants) | 89 | 84 | 80 | 75 | 0 | 0
  24 hr | 4.31 [2.45 to 6.16] | -1.38 [-3.24 to 0.49] | 0.24 [-2.37 to 2.85] | -1.61 [-3.22 to -0.01] |  |
Statistical Analysis 1: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 0.5 Hr; LS Mean Difference = 0.52, 90% CI 2-sided [-1.11 to 2.14]
Statistical Analysis 2: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 1 Hr; LS Mean Difference = 0.36, 90% CI 2-sided [-1.26 to 1.98]
Statistical Analysis 3: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 2 Hr; LS Mean Difference = 1.31, 90% CI 2-sided [-1.04 to 3.66]
Statistical Analysis 4: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 3 hr; LS Mean Difference = 4.27, 90% CI 2-sided [1.90 to 6.64]
Statistical Analysis 5: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 4 Hr; LS Mean Difference = 7.00, 90% CI 2-sided [4.35 to 9.64]
Statistical Analysis 6: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 6 Hr; LS Mean Difference = 7.85, 90% CI 2-sided [4.35 to 9.64]
Statistical Analysis 7: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 8 Hr; LS Mean Difference = 9.25, 90% CI 2-sided [6.71 to 11.80]
Statistical Analysis 8: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 12 Hr; LS Mean Difference = 4.81, 90% CI 2-sided [2.27 to 7.35]
Statistical Analysis 9: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 14 Hr; LS Mean Difference = 3.57, 90% CI 2-sided [0.91 to 6.23]
Statistical Analysis 10: Comparison: MK-8189 48 mg Day 1 vs Placebo Day 1; Test type: Other — LS Mean Difference 24 Hr; LS Mean Difference = 5.01, 90% CI 2-sided [3.18 to 6.85]
Statistical Analysis 11: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 1 Hr; LS Mean Difference = 3.95, 90% CI 2-sided [1.56 to 6.34]
Statistical Analysis 12: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 2 Hr; LS Mean Difference = 3.92, 90% CI 2-sided [1.49 to 6.35]
Statistical Analysis 13: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 3 Hr; LS Mean Difference = 4.68, 90% CI 2-sided [2.33 to 7.03]
Statistical Analysis 14: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 4 Hr; LS Mean Difference = 4.79, 90% CI 2-sided [2.45 to 7.12]
Statistical Analysis 15: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 8 Hr; LS Mean Difference = 4.82, 90% CI 2-sided [1.93 to 7.71]
Statistical Analysis 16: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 11 Hr; LS Mean Difference = 5.30, 90% CI 2-sided [2.51 to 8.09]
Statistical Analysis 17: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 14 Hr; LS Mean Difference = 5.85, 90% CI 2-sided [2.97 to 8.74]
Statistical Analysis 18: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 16 Hr; LS Mean Difference = 4.12, 90% CI 2-sided [1.79 to 6.45]
Statistical Analysis 19: Comparison: MK-8189 80 mg Day 2 vs Placebo Day 2; Test type: Other — LS Mean Difference 24 Hr; LS Mean Difference = 0.78, 90% CI 2-sided [-1.69 to 3.26]

5. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to ~30 days after each dose
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Days 1 and 2: Participants received placebo on Day 1 and Day 2 (data are pooled).
Arm/Group | MK-8189 48 mg Day 1 | Placebo Days 1 and 2 | MK-8189 80 mg Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 98 | 90 | 92 | 89 | 89
Participants | 25 | 16 | 21 | 7 | 11

6. Secondary Outcome: Maximum Concentration (Cmax) of MK-8189
Description: Cmax is the maximum plasma concentration of MK-8189.
Time Frame: Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 14, 24 hours postdose; Day 2: 0.5, 1, 2, 3, 4, 8, 11, 14, 16, 24, 36, 48, 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 96 | 0 | 91 | 0 | 0 | 0
nM | 1290 (50.6) |  | 2360 (52.4) |  |  |

7. Secondary Outcome: Concentration of MK-8189 at 24 Hours (C24) Post-dose
Description: C24 is the plasma concentration 24 hours postdose.
Time Frame: Day 1 and Day 2: 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-8189 48 mg Day 1 | Placebo Day 1 | MK-8189 80 mg Day 2 | Placebo Day 2 | Moxifloxacin 400 mg Day 2 | Standard Image Placebo Day 1
Number analyzed (Participants) | 91 | 0 | 86 | 0 | 0 | 0
nM | 992 (83.7) |  | 1660 (87.4) |  |  |

8. Secondary Outcome: Apparent Terminal Half-life (t½) of MK-8189
Description: t½ is the time required for the Cmax plasma concentration to reduce by 50%. Per protocol, t½ was determined only for MK-8189 80 mg.
Time Frame: Day 2: 0.5, 1, 2, 3, 4, 8, 11, 14, 16, 24, 36, 48, 72 hours postdose
Population: All participants who received MK-8189 80 mg, had sufficient terminal phase data, and who complied with the protocol sufficiently to ensure that generated data will likely exhibit the effects of treatment (according to the underlying scientific model), are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- MK-8189 48 mg: Participants received a single dose of MK-8189 48 mg.
- MK-8189 80 mg: Participants received a single dose of MK-8189 80 mg.
- Moxifloxacin 400 mg: Participants received a single dose of moxifloxacin 400 mg.
- Placebo: Participants received a single dose of placebo.
Arm/Group | MK-8189 48 mg | MK-8189 80 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 0 | 85 | 0 | 0
hours |  | 9.89 (29.2) |  |

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8189
Description: Tmax is defined as the time to reach Cmax.
Time Frame: Day 1: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 14, and 24 hours postdose; Day 2: 0.5, 1, 2, 3, 4, 8, 11, 14, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | MK-8189 48 mg | MK-8189 80 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 96 | 91 | 0 | 0
hours | 14.08 [6.13 to 25.42] | 14.13 [0.00 to 35.95] |  |

10. Primary Outcome: Number of Participants Discontinuing Study Therapy Due to AE
Description: as for outcome 5
Time Frame: Up to ~30 days after each dose
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8189 48 mg Day 1 | Placebo Days 1 and 2 | MK-8189 80 mg Day 2 | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
Number analyzed (Participants) | 98 | 90 | 92 | 89 | 89
Participants | 3 | 1 | 4 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to ~30 days after each dose
Description: All treated participants are included. Treatments were administered on Day 1 and Day 2.
Groups:
- MK-8189 48 mg: Participants received a single dose of MK-8189 48 mg on Day 1.
- MK-8189 80 mg: Participants received a single dose of MK-8189 80 mg on Day 2.
- MK-8189 Placebo: Participants received placebo on Day 1 and Day 2.
Arm/Group | MK-8189 48 mg | MK-8189 80 mg | MK-8189 Placebo | Standard Image Placebo Day 1 | Moxifloxacin 400 mg Day 2
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/92 | 0/90 | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/92 | 1/90 | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 24/98 | 21/92 | 15/90 | 7/89 | 11/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-8189 48 mg (N=98) | MK-8189 80 mg (N=92) | MK-8189 Placebo (N=90) | Standard Image Placebo Day 1 (N=89) | Moxifloxacin 400 mg Day 2 (N=89)
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-8189 48 mg (N=98) | MK-8189 80 mg (N=92) | MK-8189 Placebo (N=90) | Standard Image Placebo Day 1 (N=89) | Moxifloxacin 400 mg Day 2 (N=89)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Excessive eye blinking (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Application site injury (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 2 | 0 | 0 | 0
Medical device site irritation (General disorders) | 1 | 0 | 1 | 1 | 0
Withdrawal Syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0
Orthostatic heart rate response increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 3 | 4 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 5 | 1 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 5 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Oromandibular dystonia (Nervous system disorders) | 3 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 — For standard image placebo event was presyncope (not syncope)
Tardive dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Schizoprenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0
Hallucinations auditory (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT05893862/Prot_SAP_000.pdf